CLINICAL TRIAL: NCT03121924
Title: Effect of Timing of Oocyte Denudation Before ICSI and Its Results in an Oocyte Donation Model: a Cluster Randomized Controlled Clinical Trial
Brief Title: Effect of Timing of Oocyte Denudation Before ICSI in an Oocyte Donation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2500
Record Dates: First submitted 2016-09-27; First posted 2017-04-20 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2019-08

CONDITIONS: Fertility
Keywords: oocyte denudation; preincubation; icsi; oocyte donation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediately oocyte denudation (Experimental): After the retrieval , sybling oocytes were assigned to one o more recipient and then ,the oocytes were randomized in two arms .
  The first arm is the immediately denudation and immediately ICSI of the oocytes, and in the second arm the oocyte are denuded and injected after 4 hours from the pick up .
  Interventions: Procedure: timing for oocyte denudation and Intracytoplasmatic Sperm injection
- Delayed oocyte denudation (Experimental): After the retrieval , sybling oocytes were assigned to one o more recipient and then ,the oocytes were randomized in two arms .
  In this arm, the oocyte are denuded and injected after 4 hours from the pick up .
  Interventions: Procedure: timing for oocyte denudation and Intracytoplasmatic Sperm injection

INTERVENTIONS:
Procedure: timing for oocyte denudation and Intracytoplasmatic Sperm injection — Donated oocytes were randomly allocated to two groups concerning the time of cumulus corona removal.
  The first group: After oocyte retrieval, cumulus cells were immediately removed and then ICSI was performed; in the second group, the oocyte-cumulus complexes were incubated for 4 hours. Afterwards, the granulosa cells were removedand ICSI was immediately performed.
  Other Names: cumulus corona removed; granulosa cells removed

SUMMARY:
Analyze the effect of preincubation time of oocyte on the results of ICSI in a oocyte donation model.

DETAILED DESCRIPTION:
There is an intense communication inside the follicular structure. Bidirectional information between the oocyte and the granulosa cells is needed for a normal follicular development and oocyte competence.

There are conflicting results on the effect of pre-incubation time in ICSI.

It is not clear the proper time to denudate the oocyte from the somatic cells prior to ICSI, and some authors describe a negative impact of the premature cummulus removal on the ICSI results.

The aim of this study is to investigate wheter a preincubation time between oocyte retireval and injection has any effect on the ICSI ( intracytoplasmatic sperm injection) results .

ELIGIBILITY:
Inclusion Criteria:

* Oocytes retrieved from healthy donors, younger than 32 years old , with proven maternity(preference), who meet the admission criteria of ovodonation program:
* The oocytes included will be the product of antagonist stimulation protocol and with Gnrh agonists trigger. (see annex)
* Healthy women under 50 years of age , who meet the criteria as receptors into the ovodonation program.
* Oocytes retrieved after 36.5 h + -1 h of administration of triptorelin acetate.
* Only mature oocytes, in stage MII, will be included and injected.
* Use of fresh or thawed semen for the ICSI.

Exclusion Criteria:

* Cases of severe male factor such as azoospermia or severe oligo-astheno-teratospermia( alone or combinated)
* Sperm samples from surgical procedures (biopsy / testicular or epididymal puncture)
* Donors with a polycystic ovarian profile, according to The Androgen Excess and PCOS Society (AES), 2006.
* Thawed donated oocytes
* Oocytes from patients who have previously donated within a period of less than three months.
* Donors whith poor response (oocyte retrieved less than < 4 oocytes).
* Suspicion or signs of Endometriosis in donor patient.

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 375 (Actual)
Dates: Start 2015-12-01; Primary Completion 2018-12-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Number of M2 oocytes at injection | four hours after oocyte retrieval
  Asessment of the number of M2 oocytes was made after the oocyte denudation and ICSI
Number of normal fertilized oocytes after ICSI | 24 hours
  Asessment of the normal fertilization rate was made 24 hours after the intervention.
Number of cleaving embryos | 72 hours
  The embryo cleavage was evaluated after 48 hours and 72 hours after the ICSI was performed.
Number of TOP embryos | 72 hours
  The embryos were morfologically classified into 4 categories . It considered TOP embryos those correctly fertilized at day 1, and with regular 6 to 8 cells at day 2 with less than 20% fragmentation and without multinuclear blastomeres.

SECONDARY OUTCOMES:
Implantation rate | 14 days after embryo trasfer
  The implantation rate was the ratio between the number of gestacional sacs and the number of transferred embryos.
Clinical pregnancy rate | 6 to 7 week
  Clinical pregnancy is confirmed by ultrasonography ,when one or more gestational sacs with heart activity are seen.

CONTACTS AND LOCATIONS:
Overall Officials: Romina I Pesce, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison KL, Wilson LM, Breen TM, Pope AK, Cummins JM, Hennessey JF. Fertilization of human oocytes in relation to varying delay before insemination. Fertil Steril. 1988 Aug;50(2):294-7. doi: 10.1016/s0015-0282(16)60076-6. PMID 3294045
- [Background] Jacobs M, Stolwijk AM, Wetzels AM. The effect of insemination/injection time on the results of IVF and ICSI. Hum Reprod. 2001 Aug;16(8):1708-13. doi: 10.1093/humrep/16.8.1708. PMID 11473969
- [Result] Rienzi L, Ubaldi F, Anniballo R, Cerulo G, Greco E. Preincubation of human oocytes may improve fertilization and embryo quality after intracytoplasmic sperm injection. Hum Reprod. 1998 Apr;13(4):1014-9. doi: 10.1093/humrep/13.4.1014. PMID 9619563
- [Result] Van de Velde H, De Vos A, Joris H, Nagy ZP, Van Steirteghem AC. Effect of timing of oocyte denudation and micro-injection on survival, fertilization and embryo quality after intracytoplasmic sperm injection. Hum Reprod. 1998 Nov;13(11):3160-4. doi: 10.1093/humrep/13.11.3160. PMID 9853875
- [Result] Yanagida K, Yazawa H, Katayose H, Suzuki K, Hoshi K, Sato A. Influence of oocyte preincubation time on fertilization after intracytoplasmic sperm injection. Hum Reprod. 1998 Aug;13(8):2223-6. doi: 10.1093/humrep/13.8.2223. PMID 9756300
- [Result] Ho JY, Chen MJ, Yi YC, Guu HF, Ho ES. The effect of preincubation period of oocytes on nuclear maturity, fertilization rate, embryo quality, and pregnancy outcome in IVF and ICSI. J Assist Reprod Genet. 2003 Sep;20(9):358-64. doi: 10.1023/a:1025476910771. PMID 14531646
- [Result] Hassan HA. Cumulus cell contribution to cytoplasmic maturation and oocyte developmental competence in vitro. J Assist Reprod Genet. 2001 Oct;18(10):539-43. doi: 10.1023/a:1011901923261. PMID 11699125